CLINICAL TRIAL: NCT02604589
Title: Prime "Rib" Time: Randomized Control Trial Evaluating the Use of Continuous Intercostal Nerve Blockade for Traumatic Rib Fractures
Brief Title: Continuous Intercostal Nerve Blockade for Traumatic Rib Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: resource reallocation
Sponsor: Anthony Iacco (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Anthony Iacco, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-233
Record Dates: First submitted 2015-11-02; First posted 2015-11-13 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Rib Fractures
Keywords: Catheters, Indwelling; Infusion Pumps; Anesthesia, Local; Analgesia, Patient-Controlled; Bupivacaine
MeSH Terms: conditions — Rib Fractures; Agnosia | interventions — Hydromorphone; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PCA only (Placebo Comparator): Procedure: Standard of care - Intravenous Patient Controlled Anesthesia (PCA) 0.1 mg hydromorphone hydrochloride, every 6 minutes. Boluses of 0.1 mg IV hydromorphone for uncontrolled pain up to a maximum of 2.5 mg/hr.
  Interventions: Drug: hydromorphone hydrochloride
- Bupivicaine 0.25% (LOW DOSE) (Experimental): Standard PCA infusion 0.1 mg hydromorphone hydrochloride, every 6 minutes. Bolus 0.1 mg hydromorphone for uncontrolled pain up to a maximum of 2.5 mg/hr.
  Infusion catheter placement. Bupivacaine 0.25% 4 ml/hr total for dual chamber catheter.
  Interventions: Drug: hydromorphone hydrochloride; Procedure: Infusion catheter placement; Drug: bupivicaine 0.25%
- Bupivicaine 0.5% (HIGH DOSE) (Experimental): Standard PCA infusion 0.1 mg hydromorphone hydrochloride, every 6 minutes. Bolus 0.1 mg hydromorphone for uncontrolled pain up to a maximum of 2.5 mg/hr.
  Infusion catheter placement. Bupivacaine 0.5% 4 ml/hr total for dual chamber catheter.
  Interventions: Drug: hydromorphone hydrochloride; Procedure: Infusion catheter placement; Drug: bupivicaine 0.5%

INTERVENTIONS:
Drug: hydromorphone hydrochloride — Patient-controlled narcotic analgesia pump
  Other Names: Dilaudid
Procedure: Infusion catheter placement — Placement of continuous infusion catheter and elastomeric pump into extrathoracic paraspinous space
  Other Names: OnQ pump placement
  Arms: Bupivicaine 0.25% (LOW DOSE); Bupivicaine 0.5% (HIGH DOSE)
Drug: bupivicaine 0.25% — Low Dose analgesia
  Other Names: Marciane
  Arms: Bupivicaine 0.25% (LOW DOSE)
Drug: bupivicaine 0.5% — High dose analgesia
  Other Names: Marcaine
  Arms: Bupivicaine 0.5% (HIGH DOSE)

SUMMARY:
Rib fractures are common injuries in accident patients and can be associated with significant pain during recovery. If poorly controlled, pain from splinting due to rib fractures can result in difficulty in breathing leading to incomplete expansion of lung, and even the need to put a patient on a ventilator to help them breathe. Therefore, pain control is critical in managing patients with rib fractures. To date, many studies have shown the effectiveness of continuous intercostal nerve blockade (a slow release of pain medications at the site of injury that prevents the transmission of pain signals). This approach has never been studied in a randomized fashion in rib fracture patients, and has never been compared to patient-controlled narcotic pain medication, commonly used at many hospitals. The purpose of this study is to evaluate the effectiveness of the placement of an elastomeric infusion pump (a small, external, wearable balloon used to deliver medication over time) attached to a continuous infusion catheter or "soaker" catheter (a tube which releases the pain medication through tiny holes in it, right at the site of injury) to deliver local anesthetic medication to reduce pain caused by two or more rib fractures.

DETAILED DESCRIPTION:
Treatment of rib fractures using an elastomeric infusion pump (a small, external, wearable balloon used to deliver medication over time) containing pain medication and a continuous infusion catheter or "soaker" catheter (a tube which releases the pain medication through tiny holes in it, right at the site of injury) placed in the extrathoracic paraspinous space (a site in the back that is near the broken ribs) to create a continuous intercostal nerve block is relatively novel. Truitt and colleagues have published two studies evaluating the effectiveness of this approach. A pilot study on 30 patients was published in 2010 showing that placement of these catheters was a safe, viable and effective procedure, and resulted in decreased pain scores in rib fracture patients. A second study included 102 patients studied prospectively (from the time of admission to the hospital) comparing epidural anesthesia (an injection of anesthetic into the spine) with local catheter delivery in a non-randomized fashion in 2011. This approach is beginning to be more widely used, but has never been studied in a randomized fashion, and has never been compared to patient-controlled analgesia (PCA, delivery of a pain medication by the push of a button), commonly used at many hospitals.

We hypothesize that accident patients with two or more rib fractures who receive pain control through the continuous infusion system will achieve improved pain control in a dose-dependent fashion, improved lung function, and therefore, will require less narcotic pain medication, achieve discharge criteria earlier and have a shorter hospital length of stay in comparison to patients treated with PCA alone.

ELIGIBILITY:
Inclusion Criteria:

* Admission to trauma service at Beaumont Hospital, Royal Oak, Michigan
* Two or more rib fractures in an anatomic pattern feasible for nerve blockade (unilateral or bilateral)
* Age greater than or equal to 18 years
* Ability to comprehend and endorse an informed consent

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients intubated before placement of continuous infusion catheter
* Any significant concomitant injuries potentially confounding for evaluation of the effectiveness of analgesia (eg., traumatic brain injury)
* History of an allergic reaction to local anesthetic
* Use of other regional anesthetics before evaluation (epidural or paravertebral nerve blockade)
* International Normalized Ratio (INR) > 2.0
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Iacco, MD, Principal Investigator — Beaumont Hospital, Royal Oak MI
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivicaine 0.25% (LOW DOSE): bupivicaine 0.25%: Low Dose analgesia
  Standard PCA infusion 0.1 mg hydromorphone hydrochloride, every 6 minutes. Bolus 0.1 mg hydromorphone for uncontrolled pain up to a maximum of 2.5 mg/hr.
  PLUS Infusion catheter placement. Bupivacaine 0.25% 4 ml/hr total for dual chamber catheter.
- Bupivicaine 0.5% (HIGH DOSE): bupivicaine 0.5%: High dose analgesia
  Standard PCA infusion 0.1 mg hydromorphone hydrochloride, every 6 minutes. Bolus 0.1 mg hydromorphone for uncontrolled pain up to a maximum of 2.5 mg/hr.
  PLUS Infusion catheter placement. Bupivacaine 0.5% 4 ml/hr total for dual chamber catheter.
Period: Overall Study
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Started | 3 | 5 | 2
Completed | 3 | 5 | 1
Not Completed | 0 | 0 | 1
Not completed — catheter dislodgement | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE) | Total
Number analyzed (Participants) | 3 | 5 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 6
  >=65 years | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (16.56) | 60.40 (24.93) | 63.50 (6.36) | 61.40 (18.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 6
  Male | 0 | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 2 | 10
Number of Ribs Fractured [Mean (Standard Deviation); unit: ribs] | 4.7 (2.5) | 6.6 (3.7) | 5.0 (1.4) | 5.7 (2.9)
Admission Incentive Spirometry (IS) Volume [Mean (Standard Deviation); unit: cc] — Maximal inspiratory lung volume measured by incentive spirometer (IS)
  cc | 978 (563) | 783 (630) | 1567 (818) | 998 (696)
Admission Pain Score [Median (Full Range); unit: units on a scale] — Analog pain scale of 1-10, where 1= no pain and 10= worst pain ever
  units on a scale | 8 [8 to 8] | 8 [7 to 10] | 7 [6 to 9] | 8 [6 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Use
Description: Quantity of systemic narcotic used (hydromorphone hydrochloride, Dilaudid) averaged per day over the length of hospital stay, in mg/24 hours.
Time Frame: 3 days or hospital length of stay, if less than 3 days
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group
Measure: Mean (Standard Deviation); unit: mg/24 hours over days 1-3
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
mg/24 hours over days 1-3 | 3.7 (3.5) | 8.2 (5.16) | 2.5 (0)

2. Secondary Outcome: Time to Improvement in Pulmonary Function
Description: Determine the impact of catheter-infused medications on maximal inspiratory lung volume measured by incentive spirometer (IS) as a change from baseline at 24, 48, 72 hours and at 3 days post catheter placement or at discharge (or PCA placement in comparator group). Endpoint will be the time to improvement of vital capacity to greater than 1.4 liters (or 15 mL/kg).
Time Frame: 3 days or hospital length of stay, if less than 3 days
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group. This leaves only one member to analyze; therefore standard deviation = 0.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
days | 1.7 (1.5) | 1.8 (1.6) | 1.0 (0)

3. Secondary Outcome: Time to Improvement in Pain Intensity
Description: Determine the impact of catheter-infused medications on self-reported pain intensity reported as a change from baseline (admission) at 24, 48, 72 hours and at 3 days post catheter placement or at discharge (or PCA placement in comparator group) on a 0-10 point Likert scale, with 0=no pain, and 10= the worst pain ever. Response will be defined as time to a decrease of at least two points on the scale.
Time Frame: 3 days or hospital length of stay, if less than 3 days
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group. Only one subject remains to be analyzed in that group so standard deviation = 0
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
days | 2.0 (0) | 3.0 (0) | 1.0 (0)

4. Secondary Outcome: Morbidity
Description: Collection of complications observed at any point during the hospital admission that included randomization, including pneumothorax, hemothorax, acute respiratory distress syndrome, pneumonia, empyema, need for tracheostomy, need for mechanical ventilation, length of time on mechanical ventilation, and an assessment of the degree of association of each event with the catheter insertion procedure or with underlying trauma. Each of these outcomes will be scored as yes/no.
Time Frame: 3 days or hospital length of stay, whichever is longer
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group
Measure: Number; unit: number of complications
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
number of complications | 0 | 0 | 0

5. Secondary Outcome: Mortality
Description: All cause death, death associated with infusion catheter, within 30 days from date of randomization. This outcome will be scored as yes/no and cause of death will be collected.
Time Frame: 30 days
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group
Measure: Count of Participants; unit: Participants
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
Participants | 0 | 0 | 0

6. Secondary Outcome: Hospital Length of Stay
Description: Integer days of inpatient admission in the hospital stay that included randomization.
Time Frame: from randomization to discharge, usually within the range of 5-15 days
Population: One subject withdrawn in Bupivicaine 0.5% (HIGH DOSE) group. This leaves only one subject to analyze, so standard deviation =0
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 3 | 5 | 1
days | 5.0 (2.1) | 11.1 (8.6) | 3.6 (0)

7. Secondary Outcome: Surgical Intensive Care Unit (SICU) Length of Stay
Description: Integer days of admission to the surgical intensive care unit. For patients not requiring admission to surgical intensive care, patient is not analyzed. Usual range is 3-5 days.
Time Frame: from admission to Surgical Intensive Care unit to discharge from Surgical Intensive Care Unit
Population: Only patients analyzed who had surgical intensive care unit admission.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Number analyzed (Participants) | 1 | 3 | 0
days | 2.3 (0) | 5.1 (3.4) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through the first 3 days of hospitalization.
Description: An assessment of medical records and case report forms were examined for Adverse Events or Serious Adverse Events. Reports were reviewed by the PI for accuracy and relation to study intervention.
Arm/Group | PCA Only | Bupivicaine 0.25% (LOW DOSE) | Bupivicaine 0.5% (HIGH DOSE)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCA Only (N=3) | Bupivicaine 0.25% (LOW DOSE) (N=5) | Bupivicaine 0.5% (HIGH DOSE) (N=1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Low urine output (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes